CLINICAL TRIAL: NCT05981911
Title: a Non-randomized, Prospective, Open-label Registry to Compare the Effectiveness and Safety of XIENCE Skypoint™ Stents Versus Other DESs in Patients With Coronary Artery Disease
Brief Title: Evaluation of Effectiveness and Safety of Xience Skypoint Stents in Routine Clinical Practice
Acronym: IRIS Skypoint
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Department of Cardiology, University of Ulsan College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2023-04
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stent; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- XIENCE Skypoint™ stent: Patients receiving Xience-Skypoint™ stents
  Interventions: Device: XIENCE Skypoint™ stent

INTERVENTIONS:
Device: XIENCE Skypoint™ stent — Percutaneous coronary intervention with Xience-Skypoint™ stent

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of XIENCE Skypoint stents in comparison to other drug-eluting stents (DES) in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 19 years old
2. Patients receiving Xience-Skypoint™ stents.
3. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Patients with a mixture of other DESs
2. Terminal illness with life expectancy <1 year
3. Patients with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Xience-Skypoint™ stents.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the composite event rate of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months
  the composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) at 12 months post procedure.
  A composite endpoint is an endpoint that is a combination of multiple clinical endpoints. An event is considered to have occurred if any one of several different events is observed.

SECONDARY OUTCOMES:
the event rate of all cause death | 5 years
the event rate of cardiac death | 5 years
the event rate of nonfatal myocardial infarction | 5 years
the composite event rate of death, or nonfatal myocardial infarction (MI) | 5 years
the composite event rate of cardiac death, or nonfatal myocardial infarction (MI) | 5 years
the event rate of Target- Vessel Revascularization (TVR) | 5 years
the event rate of Target- lesion Revascularization (TLR) | 5 years
the event rate of stent thrombosis | 5 years
  according to an Academic Research Consortium (ARC) criteria
the event rate of stroke | 5 years
the event rate of Procedural success | 7 days
  (defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided